CLINICAL TRIAL: NCT04187755
Title: Cefepime vs Ceftazidime as Empirical Therapy for Neutropenic Fever in Pediatric Acute Leukemia: Review of Temperature and Absolute Neutrophil
Brief Title: Cefepime vs Ceftazidime as Empirical Therapy for Neutropenic Fever
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Murti Andriastuti, Doctor, Doctor, Study director, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CefepimevsCeftazidime
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Neutropenia, Febrile; Leukemia; Pediatric Cancer; Antibiotic Reaction
Keywords: fever; neutropenia; temperature; absolute neutrophil count; antibiotic
MeSH Terms: conditions — Febrile Neutropenia; Leukemia; Neoplasms; Fever; Neutropenia | interventions — Ceftazidime; Cefepime

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into two intervention groups, ceftazidime and cefepime, each group consist of 36 patients. Patients were treated, the results were noted after 72 hours.
Who Masked: Investigator
Masking Description: This study is a randomized controlled trial with single blinding, participants were assigned into ceftazidime and cefepime group. Investigator did not know the randomization done by the other party
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Participants were given ceftazidime as the antibiotic therapy with standard regimens and dose of antibiotic
  Interventions: Drug: Ceftazidime Injection
- Group II (Experimental): Participants were given cefepime as the antibiotic therapy with standard regimens and dose of antibiotic
  Interventions: Drug: Cefepime Injection

INTERVENTIONS:
Drug: Ceftazidime Injection — Ceftazidime was administered intravenously with usual standard dose for serious infection (50 mg/kgBW/dose, 6 hourly)
  Arms: Group I
Drug: Cefepime Injection — Cefepime was administered intravenously with usual standard dose for serious infection (50 mg/kgBW/dose, 8 hourly)
  Arms: Group II

SUMMARY:
Empirical antibiotic therapy has been known to reduce the mortality and morbidity rate in neutropenic fever. Until now, ceftazidime was the first line choice of neutropenic fever. However, resistance against ceftazidime has been reported. Several countries have reported cefepime in reducing fever and shorten the length of hospitalization better than ceftazidime. This study is aimed to compare the effectivity of ceftazidime and cefepime to reduce fever and to increase the absolute neutrophils count (ANC) in the first 72 hours.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with single blinding, conducted in the children's hematology-oncology wards of Cipto Mangunkusumo Hospital and Harapan Kita Children's Hospital in Jakarta, December 2018 through May 2019. Study population includes all children with leukemia with febrile neutropenia episodes that are being hospitalized in our hospitals in the appropriate time. Subjects were chosen by consecutive sampling. Inclusion criteria includes children with leukemia aged 1 month to 18 years old undergoing chemotherapy, having fever of ≥ 38,3 degree celsius in axillar temperature with ANC < 1000/mm3. Patients' parents or guardians must be willing to participate and willing to sign a written informed consent form. Exclusion criteria includes patients with a history of penicillin or cephalosporin allergy and/or patients with kidney dysfunction. Block randomization was done to place each patient into cefepime or ceftazidime group. Data analysis was done using SPSS ver. 21 software. Numerical data was shown as mean with standard deviation if the data is normally distributed or median with minimum-maximum value if the data is not normally distributed. Chi-square as the correlation test was done in order to determine the association between free and dependent variables, based on nominal data. Mann Whitney test was done as the correlation test in order to test the difference between medians of uncoupled groups and one categorical variable, and one interval variable and the not normally distributed data.

ELIGIBILITY:
Inclusion Criteria:

* children with leukemia aged 1 month to 18 years old undergoing chemotherapy
* having fever of ≥ 38,3 0C in axillar temperature
* ANC < 1000/mm3
* patients' parents or guardians must be willing to participate and willing to sign a written informed consent form

Exclusion Criteria:

* patients with a history of penicillin or cephalosporin allergy
* patients with kidney dysfunction

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Temperature decrease | after 72 hours of antibiotic adminstration
  Decrease of temperature <= 37,5 degree celsius after administration of antibiotic
Increase of Absolute Neutrophil Count | after 72 hours of antibiotic administration
  ANC >= 1000

CONTACTS AND LOCATIONS:
Overall Officials: Murti A MD,PhD, Study Director — Indonesia University
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided